CLINICAL TRIAL: NCT01585740
Title: Effect of Ringer's Lactate on Maternal and Neonatal pH in Caesarean Section at Mulago Hospital, a Randomized Trial
Brief Title: Ringer's Lactate Versus Normal Saline in Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Principal Investigator, Faculty of Medicine, Dr. Emmanuel Timarwa Ayebale, Makerere University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FluidObs-1
Record Dates: First submitted 2012-04-05; First posted 2012-04-26 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Normal Anion Gap Metabolic Acidosis
Keywords: Hyperchloraemic metabolic acidosis; Neonatal acidosis; Neonatal hyperchloraemia; Base excess; Metabolic acidosis; Caesarean section; Normal saline; Ringer's Lactate; Postoperative morbidity
MeSH Terms: conditions — Acidosis | interventions — Saline Solution; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal Saline (Active Comparator): 250 patients in this arm assigned to receive normal saline as the study fluid
  Interventions: Drug: 0.9% Normal Saline
- Ringer's Lactate (Active Comparator): 250 patients in this arm assigned to receive Ringer's Lactate as the study fluid
  Interventions: Drug: Ringer's Lactate

INTERVENTIONS:
Drug: 0.9% Normal Saline — Crystalloid fluid
  Other Names: Normal saline
  Arms: Normal Saline
Drug: Ringer's Lactate — Crystalloid fluid
  Other Names: Lactated Ringer's; Hartmann's Solution
  Arms: Ringer's Lactate

SUMMARY:
The objective of this study is to compare the effect on mean maternal and neonatal pH, and 24-hour postoperative morbidity, following intraoperative infusion of Ringer's Lactated versus normal saline in caesarean section at Mulago Hospital.

The null hypothesis is that intraoperative infusion of Ringer's Lactate in caesarean section at Mulago Hospital will not result in 30% less mean maternal and neonatal pH change than intraoperative infusion of normal saline.

DETAILED DESCRIPTION:
Fluid therapy in caesarean section surgery in Mulago Hospital is done mostly with 0.9% normal saline (NS). Several studies have highlighted the complications associated with large infusion of normal saline. Few studies have compared the effects of an alternative crystalloid, Ringer's Lactate (RL), on perinatal pH and postoperative morbidity in caesarean section surgery.

This trial will be performed in Mulago Hospital Labour Ward theatre on parturients who consent and are scheduled for either elective or emergency caesarean section under spinal anaesthesia from September 2011 to May 2012. Study fluid will be administered intraoperatively only. Preoperative and postoperative venous blood samples will be drawn for venous blood gases, serum urea and creatinine. Placental umbilical arterial cord blood will also be drawn for neonatal arterial blood gases. Mothers will be followed up for 24 hours for incidence of postoperative morbidity.

ELIGIBILITY:
Inclusion Criteria:

* All parturients who consent for the study.
* Up to American Society of Anesthesiology (ASA) class ІІ/E.

Exclusion Criteria:

* Failed spinal anaesthesia that has to be converted to general anaesthesia.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in Maternal pH from preoperative baseline | Intraoperatively
  The aim is to study the effect of the study fluid on maternal pH. pH will be measured preoperatively and immediately postoperatively before the patient leaves the recovery room.

SECONDARY OUTCOMES:
Neonatal pH | Within 30 seconds of umbilical cord ligature
  A sample of umbilical arterial cord blood will be drawn after ligating the cord to measure neonatal pH
Change in maternal base excess from preoperative baseline | Intraoperatively
  The aim is to study the effect of the study fluid on maternal base excess. Base excess will be measured preoperatively and immediately postoperatively before the patient leaves the recovery room.
Number of mothers with postoperative morbidity events | 24 hours postoperatively
  Using a Post-Operative Morbidity Survey (POMS) mothers will be followed up postoperatively for 24 hours assessing incidence of morbidity in the following systems: Pulmonary, Renal, Gastrointestinal, Cardiovascular, Neurological, and Hematological.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel T Ayebale, Anaesthesia, Principal Investigator — Makerere University
Locations (1):
- Mulago Hospital Labour Suite Operating Theatre, Kampala, Uganda

REFERENCES:
- [Derived] Ayebale ET, Kwizera A, Mijumbi C, Kizito S, Roche AM. Ringer's Lactate Versus Normal Saline in Urgent Cesarean Delivery in a Resource-Limited Setting: A Pragmatic Clinical Trial. Anesth Analg. 2017 Aug;125(2):533-539. doi: 10.1213/ANE.0000000000002229. PMID 28682955